CLINICAL TRIAL: NCT00098813
Title: A Phase II Study of Single Agent Depsipeptide (FK228) in Radioiodine (RAI)-Refractory Metastatic Non-medullary (Papillary, Follicular, and Hurthle Cell Variants) Thyroid Carcinoma
Brief Title: Romidepsin in Treating Patients With Recurrent and/or Metastatic Thyroid Cancer That Has Not Responded to Radioactive Iodine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01458; 04-059; N01CM62206 (NIH); CDR0000396783 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Thyroid Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — romidepsin; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis; Procedure: positron emission tomography

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase II trial is studying how well romidepsin works in treating patients with recurrent and/or metastatic thyroid cancer that has not responded to radioactive iodine. Romidepsin may stop the growth of tumor cells by blocking the some of the enzymes needed for cell growth. It may also help radioactive iodine and chemotherapy work better by making tumor cells more sensitive to the drug

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of romidepsin (depsipeptide), in terms of the proportion of patients achieving a complete or partial response or disease stabilization, in patients with progressive recurrent and/or metastatic non-medullary thyroid carcinoma that is refractory to radioactive iodine (RAI).

II. Determine the safety and tolerability of this drug in these patients.

SECONDARY OBJECTIVES:

I. Document changes in RAI uptake by comparing pre- and post-treatment RAI scans in patients treated with this drug.

II. Evaluate changes in the expression of the Na+/I- symporter (NIS) in tumors, as measured by immunohistochemistry on pre- and post-treatment biopsy specimens; and real time reverse transcriptase polymerase chain reaction (RT-PCR) for NIS mRNA on pre- and post-treatment changes biopsy specimens.

III. Determine post-treatment changes in serum thyroglobulin in patients treated with this drug.

IV. Correlate changes in post-treatment positron-emission tomography scans with whole-body RAI scans in patients treated with this drug.

OUTLINE:

Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-medullary thyroid carcinoma, including the following cell types:

  * Papillary
  * Follicular
  * Variants of papillary or follicular
  * Hürthle cell
* Recurrent and/or metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Progressive disease during or after prior treatment, as defined by >= 1 of the following criteria:

  * Presence of new or progressive lesions on CT scan or MRI
  * New lesions on bone or positron-emission tomography scan
  * Rising thyroglobulin level

    * Minimum of 3 consecutive rises with an interval of >= 1 week between each determination
* Refractory to radioactive iodine (RAI)

  * Absent or insufficient RAI-uptake documented by whole-body RAI scan within the past 6 months

    * At least 1 lesion with absent RAI-uptake required for insufficient uptake
* No known brain metastases
* Performance status - Karnofsky 60-100%
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,00/mm^3
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Chronic active viral hepatitis allowed provided patient is clinically stable and fulfills liver function eligibility criteria
* Creatinine normal
* Creatinine clearance >= 60 mL/min
* QTc =< 480 msec by ECG
* ST segment depression < 2 mm
* LVEF >= 50 % by echocardiogram
* No left ventricular hypertrophy, as defined by end-diastolic wall thickness > 12 mm in both the left ventricular posterior wall as well as septum or restrictive cardiomyopathy
* No history of any of the following cardiac diseases:

  * Canadian Cardiovascular Society (CCS) class II-IV angina pectoris
  * Myocardial infarction within the past 12 months
  * Sustained ventricular tachycardia, ventricular fibrillation, Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator
  * Any cardiac arrhythmia requiring digitalis or another antiarrhythmic medication other than a beta blocker or calcium channel blocker
  * No uncontrolled hypertension (i.e., blood pressure >= 160/95)
  * Mobitz II second degree block in patients who do not have a pacemaker

    * First degree or Mobitz I second degree block, bradyarrhythmias or sick sinus syndrome require Holter monitoring and evaluation by cardiology
  * Uncontrolled dysrhythmias
* No history of congenital long QT syndrome
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Thyroid stimulating hormone normal or suppressed
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to FR901228
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other concurrent uncontrolled illness
* At least 4 weeks since prior biologic or targeted agents (e.g., interferon alfa, thalidomide, octreotide, or cetuximab)
* No concurrent antineoplastic biologic agents
* No prior FR901228 (depsipeptide)
* No prior cytotoxic chemotherapy

  * Cytotoxic chemotherapy as a radiosensitizer allowed provided >= 3 months since prior administration
* No other concurrent antineoplastic chemotherapy
* Not specified
* At least 4 weeks since prior external beam radiation therapy

  * Documented disease progression required if patient received external beam radiotherapy to index lesions
* At least 3 months since prior RAI therapy

  * Diagnostic studies using =< 12 mCi of RAI are not considered RAI therapy
* No concurrent antineoplastic radiotherapy
* At least 2 weeks since prior anticancer cyclooxygenase-2 (COX-2) inhibitors, isotretinoin, or complementary medications
* At least 4 weeks since prior tyrosine kinase inhibitors (e.g., gefitinib or erlotinib)
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent drugs known to have histone deacetylase inhibitor activity (e.g., valproic acid)
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No concurrent hydrochlorothiazide
* No concurrent treatment dose warfarin
* No concurrent agents that cause QTc prolongation
* Concurrent daily aspirin given after myocardial infarction or COX-2 inhibitors at standard anti-inflammatory or pain doses allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, Principal Investigator — Memorial Sloan-Kettering Cancer Center at Suffolk
Locations (1):
- Memorial Sloan-Kettering Cancer Center at Suffolk, Commack, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 10/12/2004 Protocol Closed to Accrual 04/22/2008 Primary Completion Date 08/11/2009 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Treatment (Romidepsin)
Started | 20
Completed | 1
Not Completed | 19
Not completed — Death | 8
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Not completed — Progression of Disease | 1
Not completed — Other complicating disease | 1
Not completed — Reversal of RAI resistance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (34.64823228)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Tumor Major Response Rate (Including Stable Disease) as Measured by RECIST Criteria
Time Frame: From start of treatment to 8 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 11
participants
  Stable Disease | 10
  Progression of Disease | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Romidepsin)
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Romidepsin) (N=20)
AST, SGOT (Investigations) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Death-Sudden Death (General disorders) | 1 (1)
Death-Disease Progression (General disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Fistula, GI-Small bowel NOS (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decrease (Investigations) | 1 (1)
Neuropathy-motor (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1/1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Prolonged QTc interval (Investigations) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Romidepsin) (N=20)
ALT, SGPT (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hemoglobin decrease (Blood and lymphatic system disorders) | 2 (2)
White blood cell decrease (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Lymphocyte decrease (Investigations) | 7 (7)
Neutrophil count decrease (Investigations) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less